CLINICAL TRIAL: NCT06100562
Title: Dance Program for Youth With Cerebral Palsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Scottish Rite Hospital for Children (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU-2023-0893
Record Dates: First submitted 2023-10-17; First posted 2023-10-25 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Cerebral Palsy
Keywords: Dance; Action Observation
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dance Program (Experimental): 10-week adapted dance program (20 hours)
  Interventions: Behavioral: Adapted Dance Program

INTERVENTIONS:
Behavioral: Adapted Dance Program — * Participants will attend a 2x/weekly adaptive dance session for 10 weeks. If participants miss a class due to illness or an unexpected event (loss of transportation, family emergency/need) they will receive a video of the content missed and can complete the session at home.
  * Each class will start with a 10 min warm-up that will include stretching and motor games.
  * Learn a section of choreography every session using action-based intervention for 30 minutes.
  * Break for 5 min.
  * Improvisation part of class for 10 min.
  * Cool-down for 5 min.

SUMMARY:
The goal of this prospective cohort study is to learn about the impact of an adapted dance program in youth with cerebral palsy. The main questions it aims to answer are:

1. Are there clinically significant benefits for children with cerebral palsy who participate in an Adaptive Dance Program?
2. Is it feasible to implement an adaptive dance program using action-observation principles for children diagnosed with Cerebral Palsy (CP)? Participants will complete a pre-dance program assessment, participate in a 10-week dance program (20 hours), and complete a post-dance program assessment.

DETAILED DESCRIPTION:
Purpose:

Cerebral palsy (CP) is defined as a group of permanent disorders of the development of movement and posture that are attributed to non-progressive disturbances which occurred in the developing fetal or infant brain. As children with CP experience development and growth, motor disorders present along with disorders related to sensation, perception, cognition, and/or a seizure disorder. The way that CP manifests itself can change over time as a child grows and their surrounding environment changes, however, the lesion does not change. Throughout childhood and adolescence, a common obstacle that children with cerebral palsy face is a lack of participation and inclusion in the same leisure activities containing physical activity as their peers due to physical, cognitive, and social limitations. Currently, there is limited research pertaining to the concepts of adapted dance and its relation to children with CP and in turn, limited information about the benefits that these programs offer to the target population.

Background and Intervention Children with CP may not participate in the same leisure activities containing physical activity as their peers due to physical, cognitive, and social limitations. Children with CP who lack opportunities for physical activity are at increased risk for fatigue, injury, and pain secondary to maladaptation resulting from exacerbating physical impairments. To decrease these risks, it is imperative that children with CP participate in physical activity and develop a habit of healthy exercise. However, opportunities for physical activity must have accommodations for physical and cognitive deficits experienced by this population. Thus, an adapted sports program, such as dance, can be developed to cater to the target population. The program developed should be a physical activity that is meaningful and engaging. Thus, an adapted dance or sports program for the target population could be an effective solution to the obstacle.

Of the current research conducted on adaptive dance programs for children with CP, there is an overall theme of the active ingredients used in the programs. Each dance class was 60 minutes in length for 2-3x per week depending on the study. Most of the dance programs recruited volunteers to support participants throughout the dance class as needed. All programs consisted of a warm-up section and a cool-down portion at the end of class. The type of dance ranged in each study from hip-hop, ballet, and a variety of all dance types. The major theme of all adaptive dance programs for children with CP included focus on repetition of movements and an improvisation portion of the class. Dance movements were focused on balance, postural control, and directional movements. All programs consisted of a dance performance for participants' families and friends. The main outcomes from included significant gait improvement and control of movements. Major outcomes of an adaptive dance program can include significant improvement in coordination, balance, and endurance.

The use of the action-observation treatment intervention strategy has yielded a significant amount of evidence that shows the activation of the mirror neuron system can help improve specific motor skills. This motor learning technique has been successfully applied in a variety of adult populations such as stroke patients and Parkinson's disease patients, as well as more recently, children with cerebral palsy. In the context of rehabilitation sessions, patients typically work on one action per session, and this action is separated into 3 to 4 consecutive motor actions. Each action is observed for at least 3 minutes, with the total action then taking 12 minutes to observe. Actions are shown from multiple perspectives to further enhance learning. Following the observation, participants spend at least 2 minutes imitating the observed actions. The total time a session takes is typically 30 minutes.

In the context of a dance class, the research team will incorporate an action-observation technique as a method of teaching choreography steps. A section of a dance routine will be focused on for the duration of one class session, with the dance section broken up into 3 to 4 smaller movements. The environmental aspect of adding a mirror will add multiple perspectives for participants to observe the instructor performing dance actions, which could enhance learning and comprehension of dance moves.

Study Design A quasi-experimental mixed-method study will be conducted with clinical assessments completed pre-intervention and post-intervention to determine the feasibility and the impact of the intervention. The intervention will consist of participating in a 1-hour class, two times a week for 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cerebral palsy
* GMFCS levels 1 or 2
* MACS levels 1-3
* Aged 4-17 years
* Able to follow directions in English
* Ability to complete the assessment protocol
* Does not have any restrictions/contraindications following a medical procedure that prohibits movement

Exclusion Criteria:

* has uncontrolled epilepsy
* has severe behavioral problems
* unable to complete the assessment protocol

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2024-01-22 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Pediatric Balance Scale (PBS) | within 2 weeks of start of intervention (pre-intervention), within 2 weeks of end of intervention (post-intervention)
  a 14-item criterion referenced measure that tests functional balance for pediatric patients in everyday tasks with a sum score of 0-56. A higher score represents better balance.
6 minute walk test (6MWT) | within 2 weeks of start of intervention (pre-intervention), within 2 weeks of end of intervention (post-intervention)
  a standardized, self-paced walking test that is used to measure functional ability; the score is the amount of meters walked in 6 minutes; longer distances walked represents better function
The Cerebral Palsy Quality of Life Questionnaire (CPQOL) | within 2 weeks of start of intervention (pre-intervention), within 2 weeks of end of intervention (post-intervention)
  a standardized patient reported outcome measure that measures quality of life; it is completed by the caregiver and by children with CP ages 9+; each item is rated on a scale from 1-9, higher ratings indicate better quality of life
Child and Adolescent Scale of Participation (CASP) | within 2 weeks of start of intervention (pre-intervention), within 2 weeks of end of intervention (post-intervention)
  20-item caregiver questionnaire that measures a child or adolescent's participation in home, school, and community with a sum score of 20-80; a higher score represents higher participation

SECONDARY OUTCOMES:
Modified Ashworth Scale (MAS) | within 2 weeks of start of intervention (pre-intervention), within 2 weeks of end of intervention (post-intervention)
  standardized measurement of tone on a 5 point scale (0, 1, 1+, 2, 3); a higher score represents increased tone
Quality of Upper Limb Extremity Skills Test (QUEST) (optional) | within 2 weeks of start of intervention (pre-intervention), within 2 weeks of end of intervention (post-intervention)
  standardized, criterion-referenced assessment that measures dissociated movement, grasp, protective extension, and weight bearing that is reported using a standard score ranging from 0-100. A higher score represents better upper limb function.
Bruininks-Oseretsky Test of Motor Proficiency (BOT-2) -subsections (bilateral coordination and upper limb coordination) (optional) | within 2 weeks of start of intervention (pre-intervention), within 2 weeks of end of intervention (post-intervention)
  standardized, norm-referenced assessment that measures fine and gross motor skills; subtests are scored using scaled scores with a mean of 15 and standard deviation of 5. A higher score represents higher motor performance.

OTHER OUTCOMES:
Demographic information | within 2 weeks of start of intervention (pre-intervention)
  including age in years, gender, etiology of cerebral palsy, previous exposure to therapy (qualitative)
Manual Ability Classification Scale (MACS) | within 2 weeks of start of intervention (pre-intervention)
  The Manual Ability Classification Scale describes how children with cerebral palsy use their hands during activities of daily living with 1 being the least functional and 5 being the most functional
Gross Motor Function Classification System (GMFCS) | within 2 weeks of start of intervention (pre-intervention)
  The Gross Motor Function Classification Systems is a 5-level classification system that describes the gross motor function of children and youth with cerebral palsy with 1 being the lowest functioning and 5 being the highest

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Christie, MD, Principal Investigator — Scottish Rite for Children
Locations (1):
- Scottish Rite for Children, Frisco, Texas, United States

REFERENCES:
- [Background] Bax M, Goldstein M, Rosenbaum P, Leviton A, Paneth N, Dan B, Jacobsson B, Damiano D; Executive Committee for the Definition of Cerebral Palsy. Proposed definition and classification of cerebral palsy, April 2005. Dev Med Child Neurol. 2005 Aug;47(8):571-6. doi: 10.1017/s001216220500112x. PMID 16108461
- [Background] Withers JW, Muzzolon SB, Zonta MB. Influence of adapted hip-hop dancing on quality of life and social participation among children/adolescents with cerebral palsy. Arq Neuropsiquiatr. 2019 Oct 24;77(10):712-722. doi: 10.1590/0004-282X20190124. eCollection 2019. PMID 31664347
- [Background] Teixeira-Machado L, DeSantana JM. Effect of dance on lower-limb range of motion in young people with cerebral palsy: a blinded randomized controlled clinical trial. Adolesc Health Med Ther. 2019 Mar 27;10:21-28. doi: 10.2147/AHMT.S177867. eCollection 2019. PMID 30988649
- [Background] Moran Pascual P, Mortes Rosello E, Domingo Jacinto A, Belda Lois JM, Bermejo I, Medina E, Barbera Guillem R. On the Use of Dance as a Rehabilitation Approach for Children with Cerebral Palsy: A Single Case Study. Stud Health Technol Inform. 2015;217:923-8. PMID 26294586
- [Background] Owens M, Silkwood-Sherer D. Informal Dance Intervention Improves BMI and Functional Gait in an Adolescent With Cerebral Palsy: A Case Report. Pediatr Phys Ther. 2019 Oct;31(4):E26-E31. doi: 10.1097/PEP.0000000000000653. PMID 31469773
- [Background] Lopez-Ortiz C, Gaebler-Spira DJ, Mckeeman SN, Mcnish RN, Green D. Dance and rehabilitation in cerebral palsy: a systematic search and review. Dev Med Child Neurol. 2019 Apr;61(4):393-398. doi: 10.1111/dmcn.14064. Epub 2018 Oct 23. PMID 30350851